CLINICAL TRIAL: NCT04193527
Title: A Multicentre, Phase 3, Clinical Study to Compare the Striatal Uptake of a Dopamine Transporter Radioligand, DaTSCAN™ Ioflupane (123I) Injection, After Intravenous Administration to Chinese Patients With a Diagnosis of Parkinson's Disease, Multiple System Atrophy, Progressive Supranuclear Palsy, or Essential Tremor and to Healthy Controls
Brief Title: A Study to Evaluate the Diagnostic Efficacy of DaTSCAN™ Ioflupane (123I) Injection in Single Photon Emission Computed Tomography (SPECT) for the Diagnosis of Parkinsonian Syndrome (PS) in Chinese Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GE Healthcare (Industry)
Collaborators: PPD Development, LP (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GE-001-024; CTR20191992 (Registry Identifier: China Drug Evalutation)
Record Dates: First submitted 2019-12-02; First posted 2019-12-10 (Actual); Results first posted 2023-10-16 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2022-12

CONDITIONS: Parkinsonian Syndrome; Parkinson Disease(PD); Multiple System Atrophy (MSA); Progressive Supranuclear Palsy (PSP); Essential Tremor
MeSH Terms: conditions — Parkinsonian Disorders; Parkinson Disease; Multiple System Atrophy; Supranuclear Palsy, Progressive; Essential Tremor | interventions — Iodine-123; Injections; ioflupane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DaTSCAN™ ioflupane (123I) injection (Experimental): Participants with Parkinsonian Syndrome (PS), Essential Tremor (ET), and Healthy Volunteers (HV) received a single dose of DaTSCAN™ ioflupane (123I) injection. Single photon emission computed tomography (SPECT) imaging was performed between 3 to 6 hours post-injection and lasted approximately 20 minutes to 1 hour.
  Interventions: Drug: DaTSCAN™ Ioflupane (123I) Injection

INTERVENTIONS:
Drug: DaTSCAN™ Ioflupane (123I) Injection — All participants (Participants with PS, ET, and HV) received a single dose of DaTSCAN™ ioflupane (123I) injection within the range of 111 to 185 megabecquerel (MBq) (3 to 5 millicurie [mCi]) per participant at a maximum volume of 5 milliliter [mL]) intravenously on Day 1.
  Other Names: Ioflupane (123I)

SUMMARY:
This is a multicenter, open-label, non-controlled, non-randomized, phase 3 clinical study to compare the SPECT findings after a single IV administration of DaTSCAN™ ioflupane (123I) injection for patients with a clinical diagnosis of Parkinsonian syndrome (PS) involving striatal dopaminergic deficit (SDD; specifically, Parkinson's disease [PD] [SDD], multiple system atrophy [MSA] [SDD] or or progressive supranuclear palsy [PSP] [SDD]) as compared with patients with a clinical diagnosis of essential tremor (ET) (no SDD) and age-matched healthy controls.

ELIGIBILITY:
Inclusion Criteria:

For all participants:

1. Chinese male or female, aged 40 to 80 years, has agreed to sign and date the written informed consent form.

   For Healthy Volunteers:
2. Non-patient volunteers with good age-appropriate health as established by clinical examination during screening and no evidence of movement disorder by complete neurological evaluation.

   For participants with Parkinson's disease:
3. A diagnosis of clinically established or clinically probable PD in accordance with the Movement Disorder Society (MDS) Clinical Diagnostic Criteria for Parkinson's Disease.

   For participants with MSA (SDD):
4. A diagnosis of probable or possible MSA in accordance with the Second Consensus Statement on the Diagnosis of MSA.

   For participants with PSP (SDD):
5. A diagnosis of probable or possible PSP in accordance with the Clinical Criteria for the Diagnosis of Progressive Supranuclear Palsy National Institute for Neurological Disorders and Society for PSP (NINDS-SPSP)

   For participants with ET (no SDD):
6. A diagnosis of definite or probable ET in accordance with the Washington Heights-Inwood Genetic Study of Essential Tremor (WHIGET) diagnostic criteria for ET (no SDD) .

Exclusion Criteria:

1. The participant is lactating.
2. The participant is pregnant as detected by a β-human chorionic gonadotropin (β-hCG) pregnancy test.
3. A cerebral structural vascular abnormality indicative of at least 1 infarction in the region of the basal ganglia (including the internal capsule) ≥5 mm has been confirmed, preferably by magnetic resonance imaging (MRI) performed within 6 months of screening. If an MRI is not clinically feasible, cerebral CT imaging within 6 months is also acceptable.
4. The participant is diagnosed with major neurocognitive disorder by the Diagnostic and Statistical Manual of Mental Disorders (DSM) 5 criteria, or Mini-Mental State Examination total score is <24.
5. Participant is being investigated for or has been diagnosed and/or is being treated for repeated stroke with stepwise progression of Parkinson features.
6. History of repeated head injury (≥3 concussions, or history of professional sports with repeated head trauma [e.g., boxing]).
7. History of definite encephalitis (≥1 episode of confirmed encephalitis with objective residual neurologic deficit).
8. The participant is using or has insufficient washout from medication known or suspected to interact with striatal uptake through direct competition with binding of DaTSCAN™ to the dopamine transporters (i.e., amphetamine, benztropine, bupropion, cocaine, mazindol, methylphenidate, phentermine, sertraline, selective serotonin reuptake inhibitors) before the imaging visit.
9. The participant is using Chinese traditional medicine for PD treatment, which cannot be safely withdrawn for at least 1 week (7 days) before the imaging visit.
10. The participant has a moderate to severe renal impairment (e.g., serum creatinine >1.5x upper limit of normal [ULN], blood urea nitrogen [BUN] >30 mg/dL).
11. The participant has a moderate to severe hepatic impairment (bilirubin >2x ULN and alanine aminotransferase (ALT) or aspartate aminotransferase (AST)>3x ULN).
12. The participant has a history of current abuse of drugs and/or alcohol (for the previous 12 months before trial enrolment).
13. The participant has a history of occupational exposure to any radiation >50 millisievert/year (mSv/year).
14. The participant has been previously enrolled in this study or participated in a clinical study involving an investigational pharmaceutical product within 30 days prior to screening and/or any radiopharmaceutical within a minimum of 5 radioactive half-lives prior to screening.
15. The participant presents with symptoms suggestive of corticobasal degeneration or Huntington's disease.
16. The participant has known allergies to the investigational medicinal product (IMP).
17. The participant presents with any clinically active, serious, life-threatening disease with a life expectancy of less than 12 months.
18. Any laboratory value(s) exceeding the limits of normality if deemed to be clinically relevant by the investigator.
19. The participant complains of claustrophobia.
20. The participant has a moderate to severe thyroid disease (thyroid stimulating hormone [TSH] exceeding the limits of normality by more than 10%), if deemed to be clinically relevant by the investigator.

    For participants with ET:
21. The participant has at least 1 first-degree relative diagnosed with PD.

    For Healthy Volunteers:
22. History of psychiatric illness.

    For all participants:
23. It is the physician's best judgment not to include the participant in the trial.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2020-06-28 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2021-12-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- China (10):
  - Beijing Anzhen Hospital, Capital Medical University, Beijing, Chaoyang District
  - Peking Union Medical College Hospital, Beijing, Dongcheng District
  - Nanfang Hospital, Nanfang Medical Univeristy, Guangdong, Guangzhou
  - Nanjing First Hospital, Nanjing, Jiangsu
  - The Second Affilicated Hospital of Soochow University, Suzhou, Jiangsu
  - Shanghai General Hospital, Hongkou, Shanghai Municipality
  - Peking University First Hospital, Beijing
  - Beijing Friendship Hospital Afflication to Capital Medical University, Beijing
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai
  - Tianjin Medical University General Hospital, Tianjin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- DaTSCAN™ Ioflupane: Participants With Parkinsonian Syndrome (PS): Participants with PS received a single dose of DaTSCAN™ ioflupane (123I) injection within the range of 111 to 185 megabecquerel (MBq) (3 to 5 millicurie [mCi]) per participant at a maximum volume of 5 milliliter [mL] intravenously on Day 1.
- DaTSCAN™ Ioflupane: Participants With Essential Tremor (ET): Participants with ET received a single dose of DaTSCAN™ ioflupane (123I) injection within the range of 111 to 185 MBq (3 to 5 mCi) per participant at a maximum volume of 5 mL intravenously on Day 1.
- DaTSCAN™ Ioflupane: Healthy Volunteers (HV): Healthy Volunteers received a single dose of DaTSCAN™ ioflupane (123I) injection within the range of 111 to 185 MBq (3 to 5 mCi) per participant at a maximum volume of 5 mL intravenously on Day 1.
Period: Overall Study
Arm/Group | DaTSCAN™ Ioflupane: Participants With Parkinsonian Syndrome (PS) | DaTSCAN™ Ioflupane: Participants With Essential Tremor (ET) | DaTSCAN™ Ioflupane: Healthy Volunteers (HV)
Started | 75 | 75 | 22
Completed | 74 | 74 | 22
Not Completed | 1 | 1 | 0
Not completed — Other | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received an injection of Investigational Medicinal Product (IMP).
Groups:
- DaTSCAN™ Ioflupane: Participants With Parkinsonian Syndrome (PS): Participants with PS received a single dose of DaTSCAN™ ioflupane (123I) injection within the range of 111 to 185 MBq (3 to 5 mCi) per participant at a maximum volume of 5 mL intravenously on Day 1.
- DaTSCAN™ Ioflupane: Healthy Volunteer (HV): Healthy Volunteers received a single dose of DaTSCAN™ ioflupane (123I) injection within the range of 111 to 185 MBq (3 to 5 mCi) per participant at a maximum volume of 5 mL intravenously on Day 1.
- Total: Total of all reporting groups
Arm/Group | DaTSCAN™ Ioflupane: Participants With Parkinsonian Syndrome (PS) | DaTSCAN™ Ioflupane: Participants With Essential Tremor (ET) | DaTSCAN™ Ioflupane: Healthy Volunteer (HV) | Total
Number analyzed (Participants) | 75 | 75 | 22 | 172
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.0 (8.07) | 65.8 (7.24) | 61.3 (5.38) | 64.0 (7.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 38 | 14 | 86
  Male | 41 | 37 | 8 | 86
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 75 | 75 | 22 | 172
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 75 | 75 | 22 | 172
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity Analysis of the Blinded Independent Read of DaTSCAN™ SPECT Images
Description: Sensitivity was defined as positive percentage agreement and calculated as the number of true positives (TP) / (number of TP + number of false negatives [FN]): TP/(TP + FN), and a 2-sided 95% binomial confidence interval constructed around it. Only the participants with a clinical diagnosis of PS were included in the sensitivity analysis. The sensitivity of the blinded independent read of DaTSCAN™ SPECT images in detecting or excluding striatal dopaminergic deficit (SDD), when the clinical diagnosis as established by the investigator was used as the standard of truth, were summarized with by reader. Each participant's SPECT image was read by 3 blinded readers.
Time Frame: At Day 1
Population: Full-analysis set (FAS) consisted of all participants who had both a DaTSCAN™ image set and a clinical diagnosis made by the Investigator. Only the participants with a clinical diagnosis of PS were included in the sensitivity analysis.
Measure: Number (95% Confidence Interval); unit: ratio
Groups:
- DaTSCAN™ Ioflupane: Participants With Parkinsonian Syndrome (PS): Participants with PS received a single dose of DaTSCAN™ ioflupane (123I) injection within the range of 111 to 185 MBq (3 to 5 mCi per participant at a maximum volume of 5 mL) intravenously on Day 1.
Arm/Group | DaTSCAN™ Ioflupane: Participants With Parkinsonian Syndrome (PS)
Number analyzed (Participants) | 75
ratio
  Reader 1-Sensitivity | 0.851 [0.750 to 0.923]
  Reader 2-Sensitivity | 0.865 [0.765 to 0.933]
  Reader 3-Sensitivity | 0.919 [0.832 to 0.970]

2. Secondary Outcome: Normalized DaTSCAN™ Uptake Based on Region Of Interest (ROI) With Central Read (by Semi-quantitative Assessment by Use of DaTQUANT™) of DaTSCAN™ SPECT Images
Description: A semi-quantitative analysis of the striatal uptake ratios in specific regions of interest (ROIs, i.e., left and right striatum, caudate, and putamen) of DaTSCAN™ SPECT images was performed with DaTQUANT™.
Time Frame: At Day 1
Population: Full-analysis set (FAS) consisted of all participants who had both a DaTSCAN™ image set and a clinical diagnosis made by the Investigator.
Measure: Mean (Standard Deviation); unit: ratio
Groups:
- DaTSCAN™ Ioflupane: Participants With Parkinsonian Syndrome (PS): Participants with PS received a single dose of DaTSCAN™ ioflupane (123I) injection within the range of 111 to 185 megabecquerel (MBq) (3 to 5 mCi) per participant at a maximum volume of 5 mL intravenously on Day 1.
Arm/Group | DaTSCAN™ Ioflupane: Participants With Parkinsonian Syndrome (PS) | DaTSCAN™ Ioflupane: Participants With Essential Tremor (ET) | DaTSCAN™ Ioflupane: Healthy Volunteers (HV)
Number analyzed (Participants) | 75 | 75 | 22
ratio
  Anterior putamen right ratio | 1.29315 (0.577528) | 2.70530 (0.577359) | 2.94013 (0.835608)
  Anterior putamen left ratio | 1.30474 (0.635803) | 2.67536 (0.585852) | 2.92746 (0.784174)
  Caudatus asymmetry ratio | 0.10454 (0.083195) | 0.03906 (0.029737) | 0.04212 (0.023939)
  Caudatus left ratio | 1.70232 (0.758242) | 2.87229 (0.648102) | 3.05874 (0.866446)
  Caudatus right ratio | 1.71398 (0.660892) | 2.86571 (0.616034) | 2.99258 (0.885231)
  Putamen to caudatus left ratio | 0.81527 (0.113790) | 0.91598 (0.071819) | 0.94217 (0.075958)
  Putamen to caudatus right ratio | 0.80208 (0.094132) | 0.92631 (0.076093) | 0.95685 (0.060599)
  Putamen asymmetry ratio | 0.08884 (0.070714) | 0.03472 (0.026388) | 0.03066 (0.022587)
  Putamen left ratio | 1.16697 (0.578536) | 2.53527 (0.577060) | 2.80555 (0.788140)
  Posterior putamen left ratio | 0.89624 (0.506444) | 2.26000 (0.592376) | 2.56593 (0.817882)
  Posterior putamen right ratio | 0.86673 (0.514910) | 2.28143 (0.583230) | 2.53907 (0.861909)
  Putamen right ratio | 1.15783 (0.542656) | 2.57079 (0.567985) | 2.81286 (0.834213)
  Striatum asymmetry ratio | 0.09290 (0.069194) | 0.02879 (0.023420) | 0.02774 (0.019084)
  Striatum left ratio | 1.34682 (0.614929) | 2.64850 (0.584689) | 2.89059 (0.801328)
  Striatum right ratio | 1.32485 (0.560168) | 2.65936 (0.566834) | 2.86683 (0.843327)

3. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs), and Serious TEAEs
Description: An adverse event (AE) was any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this investigational product (IP) or medicinal product. A Serious Adverse Event(SAE) was any untoward medical occurrence that at any dose met one, more of the following criteria: results in death, life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent, significant disability/incapacity, a congenital abnormality/birth defect, an important medical event. A TEAE was any event emerging or manifesting at or after the initiation of treatment with an IP or medicinal product or any existing event that worsens in either intensity or frequency following exposure to the IP or medicinal product. Number of participants with TEAEs and serious TEAEs were reported.
Time Frame: From start of study drug administration up to Day 4
Population: Safety population included all participants who received an injection of Investigational Medicinal Product (IMP).
Measure: Count of Participants; unit: Participants
Groups:
- DaTSCAN™ Ioflupane: Participants With Parkinsonian Syndrome (PS): Participants with PS received a single dose of DaTSCAN™ ioflupane (123I) injection within the range of 111 to 185 MBq (3 to 5 mCi) per participant at a maximum volume of 5mL intravenously on Day 1.
Arm/Group | DaTSCAN™ Ioflupane: Participants With Parkinsonian Syndrome (PS) | DaTSCAN™ Ioflupane: Participants With Essential Tremor (ET) | DaTSCAN™ Ioflupane: Healthy Volunteers (HV)
Number analyzed (Participants) | 75 | 75 | 22
Participants
  Participants with TEAEs | 12 | 13 | 8
  Participants with Serious TEAEs | 0 | 0 | 0

4. Primary Outcome: Specificity Analysis of the Blinded Independent Read of DaTSCAN™ SPECT Images
Description: Specificity was defined as negative percentage agreement and calculated as the number of true negatives (TN) / (number of TN + number of false positives [FP]): TN/(TN + FP), and a 2-sided 95% binomial confidence interval constructed around it. For the specificity analysis, only participants with a clinical diagnosis of ET were included; the HVs were excluded from this analysis. The specificity of the blinded independent read of DaTSCAN™ SPECT images in detecting or excluding striatal dopaminergic deficit (SDD), when the clinical diagnosis as established by the investigator was used as the standard of truth, were summarized with by reader. Each participant's SPECT image was read by 3 blinded readers.
Time Frame: At Day 1
Population: Full-analysis set (FAS) consisted of all participants who had both a DaTSCAN™ image set and a clinical diagnosis made by the Investigator. Only participants with a clinical diagnosis of ET were included and the HVs were excluded from the specificity analysis.
Measure: Number (95% Confidence Interval); unit: ratio
Arm/Group | DaTSCAN™ Ioflupane: Participants With Essential Tremor (ET)
Number analyzed (Participants) | 75
ratio
  Reader 1-Specificity | 0.933 [0.851 to 0.978]
  Reader 2-Specificity | 0.960 [0.888 to 0.992]
  Reader 3-Specificity | 0.813 [0.707 to 0.894]

ADVERSE EVENTS:
Time Frame: From start of study drug administration up to Day 4
Description: Safety population included all participants who received an injection of IMP.
Groups:
- DaTSCAN™ Ioflupane: Participants With Parkinsonian Syndrome (PS): Participants with PS received a single dose of DaTSCAN™ ioflupane (123I) injection within the range of 111 to 185 MBq (3 to 5 mCi) per participant at a maximum volume of 5 milliliter [mL] intravenously on Day 1.
Arm/Group | DaTSCAN™ Ioflupane: Participants With Parkinsonian Syndrome (PS) | DaTSCAN™ Ioflupane: Participants With Essential Tremor (ET) | DaTSCAN™ Ioflupane: Healthy Volunteers (HV)
All-Cause Mortality (participants affected / at risk) | 0/75 | 0/75 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/75 | 0/75 | 0/22
Other Adverse Events (participants affected / at risk) | 12/75 | 13/75 | 8/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DaTSCAN™ Ioflupane: Participants With Parkinsonian Syndrome (PS) (N=75) | DaTSCAN™ Ioflupane: Participants With Essential Tremor (ET) (N=75) | DaTSCAN™ Ioflupane: Healthy Volunteers (HV) (N=22)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Dry eye (Eye disorders) | 0 | 1 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Injection site paraesthesia (General disorders) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 2
Conjunctivitis (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Blood glucose increased (Investigations) | 0 | 1 | 2
Blood creatine phosphokinase increased (Investigations) | 2 | 0 | 0
Protein urine present (Investigations) | 1 | 1 | 0
White blood cells urine positive (Investigations) | 0 | 2 | 0
Blood phosphorus decreased (Investigations) | 0 | 1 | 0
Neutrophil count increased (Investigations) | 1 | 0 | 0
Urinary occult blood positive (Investigations) | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 5 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-11-25): https://cdn.clinicaltrials.gov/large-docs/27/NCT04193527/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-21): https://cdn.clinicaltrials.gov/large-docs/27/NCT04193527/SAP_001.pdf